CLINICAL TRIAL: NCT01540734
Title: A Single Dose PK Study Investigating the Extent of Paracetamol Absorption From Two Sustained Release Paracetamol Formulations
Brief Title: Pharmacokinetic Study Investigating the Extent of Paracetamol Absorption From a New Formulation of Paracetamol Compared With Panadol®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A2750606
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Subjects
Keywords: paracetamol; pharmacokinetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marketed paracetamol (Active Comparator): marketed formulation
  Interventions: Drug: Marketed paracetamol
- Experimental paracetamol formulation (Experimental): Experimental formulation
  Interventions: Drug: Experimental paracetamol formulation

INTERVENTIONS:
Drug: Marketed paracetamol — Marketed formulation
  Arms: Marketed paracetamol
Drug: Experimental paracetamol formulation — Experimental formulation
  Arms: Experimental paracetamol formulation

SUMMARY:
A single dose pharmacokinetic study investigating two paracetamol formulations

ELIGIBILITY:
Inclusion Criteria:

* Good general heatlh with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination

Exclusion Criteria:

* Subject does not agree to refrain from alcohol consumption for the 10-day period prior to visit 2 and throughout the remainder of the study.
* Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
* Current (within 14 days of screening) or regular use of any prescription, over the counter drugs including paracetamol/acetaminophen, herbal medicine or drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To compare bioavailability as measured by Area under the Curve in both fed and fasted states | Visit 1 through Visit 3 (Day 13)
To assess the effect of food on extent and rate of paracetamol absorption as measured by Area Under the Curve and Cmax | Visit 1 through Visit 3 (Day 13)

SECONDARY OUTCOMES:
To assess descriptive pharmacokinetic characteristics (Tmax, T1/2, AUC, Cmax) | Visit 1 through Visit 3 (Day 13)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- MDS Pharma Services NEBRASKA, Lincoln, Nebraska, United States